CLINICAL TRIAL: NCT03542552
Title: Oral Nifedipine Versus Intravenous Magnesium Sulfate for Prevention of Preterm Labor in Symptomatic Placenta Previa: Randomized Controlled Trial.
Brief Title: Nifedipine Versus Magnesium Sulfate for Prevention of Preterm Labor in Symptomatic Placenta Previa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ramy nasser, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONIMS
Record Dates: First submitted 2018-05-19; First posted 2018-05-31 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Magnesium Sulfate; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nifidipne (Active Comparator): received oral nifedipine 10 mg every 20 minutes for three doses, followed by 10 mg orally every 6 hours
  Interventions: Drug: Nifedipine
- Magnisum sulphate (Experimental): Patients in the MgSO4 group received intravenous 6 g bolus MgSO4 20% followed by a 2 g/h infusion
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Patients received intravenous 6 g bolus MgSO4 20% followed by a 2 g/h infusion
  Arms: Magnisum sulphate
Drug: Nifedipine — received oral nifedipine 10 mg every 20 minutes for three doses, followed by 10 mg orally every 6 hours
  Arms: Nifidipne

SUMMARY:
Antepartum hemorrhage is defined as bleeding from or within the female genital tract, occurring from 28+0 weeks of pregnancy and till delivery of the fetus. it occurs in 3-5% of pregnancies and is an important cause of perinatal and maternal morbidity and mortality worldwide

DETAILED DESCRIPTION:
There are many tocolytic agents may have a role in conservative management of placenta previa such as magnesium sulfate, calcium channel blockers and β-sympathormimetics. In 2004 Sharma suggests that ritodrine hydrochloride in patients with symptomatic placenta previa tends to prolong the pregnancy and result in an increase in birth weight of the babies without causing any adverse effect on the mother and fetus

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age : between 28 weeks and 37 week's gestation
* Confirmed Placenta previa; either major or minor degrees.
* Placenta previa with preterm uterine contractions

Exclusion Criteria:

* Severe attack of bleeding requiring an immediate intervention.
* Fetal heart rates instability or non-reassuring tracing
* Intrauterine fetal death or major fetal anomalies.
* If associated with abruptio placentae
* Patients with known bleeding disorders or on anticoagulant therapy
* Patients with severe medical disorders as myasthenia gravis documented magnesium toxicity.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The duration of prolongation of gestation | 1 month
  measured from the time of enrollment to the time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046